CLINICAL TRIAL: NCT03778749
Title: The Effectiveness of Electromyographic- and Acceleromyographic-based Monitors in Diagnosing Pre-existing Train-of-four Fade in Ventilated ICU Patients
Brief Title: Electromyography and Acceleromyography in Ventilated ICU Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Application of monitoring tools seemed inappropriate in ICU patients who were ventilated during a prolonged period.
Sponsor: Onze Lieve Vrouw Hospital (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Guy CAMMU, Principal Investigator, Onze Lieve Vrouw Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018/091
Record Dates: First submitted 2018-12-12; First posted 2018-12-19 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Neuromuscular Monitoring
Keywords: train-of-four monitoring; acceleromyography; electromyography; intensive care unit

STUDY DESIGN:
Intervention Model Description: Twenty mechanically ventilated ICU patients: the investigators will compare the mean TOF% between three different measurement techniques in 20 mechanically ventilated ICU patients: 1/electromyographic neuromuscular transmission monitoring at the hand muscle - 2/acceleromyographic neuromuscular transmission monitoring at the hand muscle - 3/acceleromyographic neuromuscular transmission monitoring at the eyebrow muscle; and the investigators will determine how the three TOF% values vary in each individual patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- electromyographic NMT monitoring at the hand (Experimental): In 20 mechanically ventilated ICU patients, TOF measurements will be performed every 24 hrs, once a day, at the same time, over the 72 hrs the study will take place in the ICU.
  Interventions: Diagnostic Test: TOF measurements
- acceleromyographic NMT monitoring at the hand (Experimental): In 20 mechanically ventilated ICU patients, TOF measurements will be performed every 24 hrs, once a day, at the same time, over the 72 hrs the study will take place in the ICU.
  Interventions: Diagnostic Test: TOF measurements
- acceleromyographic NMT monitoring at the eyebrow (Experimental): In 20 mechanically ventilated ICU patients, TOF measurements will be performed every 24 hrs, once a day, at the same time, over the 72 hrs the study will take place in the ICU.
  Interventions: Diagnostic Test: TOF measurements

INTERVENTIONS:
Diagnostic Test: TOF measurements — The investigators will determine how the TOF% values vary in each individual patient, over time, in ICU.

SUMMARY:
In intensive care unit (ICU) patients who are mechanically ventilated for a longer period of time, there might be a difference in accuracy and performance of neuromuscular transmission monitoring [as measured by the train-of-four (TOF)%] due to a pre-existing TOF fade, correlated to some form of acquired muscle weakness. The investigators therefore propose to search for and compare the optimal monitoring techniques (acceleromyography vs. electromyography) and the optimal muscle monitoring site (peripheral-adductor pollicis vs. central-corrugator supercilii) in ICU patients who require prolonged mechanical ventilation.

DETAILED DESCRIPTION:
The following neuromuscular transmission monitors will be used in the study: an electromyography-based monitor (TetraGraph, Senzime AB, Uppsala, Sweden) and two devices that are the newer generation of quantitative monitoring using three-dimensional acceleromyographic technology: Stimpod (Xavant Technology, Pretoria, South Africa) and TofScan (IDmed, Marseilles, France), both of which require minimal setup for use.

The stimulation pattern of both ulnar and facial nerves will be train-of-four (TOF) delivered every 1 minute, and the mean of three consecutive measurements will be calculated as the TOF% for that patient. Patients will be tested every 24 hrs, once a day, at the same time, over the 72 hrs the study will take place in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* 18 yr. old or older
* expected to require mechanical ventilation for more than 72 hrs

Exclusion Criteria:

* degenerative neurological disease
* receive drugs interfering with NMT (e.g., aminoglycosides or magnesium)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-16 (Actual)

PRIMARY OUTCOMES:
pre-existing neuromuscular fade (TOF% <90), correlated to some form of ICU acquired muscle weakness, in ICU patients mechanically ventilated for more than 72 hrs. | 72 hours of study period in ICU
  to find whether any patients show any pre-existing neuromuscular fade or develop such weakness over the 72 hours of study period in ICU

SECONDARY OUTCOMES:
fade (TOF% <90) difference between central (corrugator supercilii) and peripheral (adductor pollicis) muscles in ICU patients who require prolonged mechanical ventilation. | 72 hours of study period in ICU
  to compare the development of fade (if any develops) between central and peripheral muscles over the 72 hours of study period in ICU

OTHER OUTCOMES:
optimal monitor for use in the ICU setting | 72 hours of study period in ICU
  to determine the TOF% repeatability of the three monitors, establishing the optimal monitor for use in the ICU setting

CONTACTS AND LOCATIONS:
Overall Officials: Guy Cammu, MD,PhD, Principal Investigator — Onze-Lieve-Vrouw Ziekenhuis, Aalst, Belgium
Locations (1):
- OLV Hospital, Aalst, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Naguib M, Brull SJ, Johnson KB. Conceptual and technical insights into the basis of neuromuscular monitoring. Anaesthesia. 2017 Jan;72 Suppl 1:16-37. doi: 10.1111/anae.13738. PMID 28044330
- [Background] Cammu G, Neyens E, Coddens J, Van Praet F, De Decker K. Postoperative residual curarisation is still an issue when weaning patients in intensive care following cardiac surgery. Anaesth Intensive Care. 2018 Nov;46(6):634-636. No abstract available. PMID 30447682